CLINICAL TRIAL: NCT01563354
Title: Multicenter 3-arm Trial to Evaluate the Efficacy and Safety of Pasireotide LAR or Everolimus Alone or in Combination in Patients With Well Differentiated Neuroendocrine Carcinoma of the Lung and Thymus - LUNA Trial
Brief Title: 3-arm Trial to Evaluate Pasireotide LAR/Everolimus Alone/in Combination in Patients With Lung/Thymus NET - LUNA Trial
Acronym: LUNA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSOM230DIC03; 2011-002872-17 (EudraCT Number)
Record Dates: First submitted 2012-03-20; First posted 2012-03-27 (Estimated); Results first posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Neuroendocrine Carcinoma of the Lung and Thymus
Keywords: neuroendocrine carcinoma; lung; thymus; pasireotide LAR; everolimus,adult,SOM230,carcinoma,lung cancer,
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — pasireotide; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pasireotide LAR (Experimental): Pasireotide long acting release (LAR) 60 mg will be administered as an intra muscular (i.m.) depot injection once every 28 days starting on Day 1
  Interventions: Drug: Pasireotide LAR
- Everolimus (Experimental): Everolimus 10 mg taken orally (p.o) once daily starting on Day 1
  Interventions: Drug: Everolimus
- Pasireotide LAR and Everolimus Combination (Experimental): Pasireotide LAR 60 mg i.m. injected once every 28 days + Everolimus 10 mg p.o. daily starting on Day 1
  Interventions: Drug: Pasireotide LAR and Everolimus Combination

INTERVENTIONS:
Drug: Pasireotide LAR — 60 mg was administered as an intra muscular depot injection once every 28 days starting at Day 1
  Other Names: SOM230
  Arms: Pasireotide LAR
Drug: Everolimus — 10 mg tables administered orally once a day
  Other Names: RAD001
  Arms: Everolimus
Drug: Pasireotide LAR and Everolimus Combination — Pasireotide LAR 60 mg i.m. injected once every 28 days + Everolimus 10 mg p.o. daily
  Other Names: SOM230 + RAD001
  Arms: Pasireotide LAR and Everolimus Combination

SUMMARY:
This was a multicenter, randomized, phase II study evaluating Everolimus or Pasireotide LAR alone or in combination in adult patients with advanced (unresectable or metastatic) neuroendocrine carcinoma of the lung and thymus

DETAILED DESCRIPTION:
This was a prospective, multicenter, randomized, open-label, 3-arm, phase II study with a single-stage design in each arm. The purpose of this study was to test the effectiveness and safety of Everolimus or Pasireotide LAR alone or in combination in adult patients with advanced (unresectable or metastatic) neuroendocrine carcinoma (typical and atypical) of the lung and thymus. It was expected that a total of 120 patients with 40 patients in each arm were to be enrolled into this study. Patients were seen weekly for one month and monthly thereafter. Radiological and biochemical response assessments were performed every 3 months.

Patients with disease control (stable disease or better) in the combination arm or monotherapy with pasireotide LAR and everolimus who had not experienced unacceptable toxicity were permitted to continue treatment in the extension phase of the study and were seen every 3 months. Patients could remain in the extension phase as long as they continued to have clinical benefit and had not fulfilled any of the study discontinuation criteria. All patients had a safety follow-up visit 56 days after last treatment dose.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed advanced well differentiated typical and atypical carcinoid tumors of the lung or thymus
* Patients of all treatment lines including naive patients could have been enrolled
* At least one measurable lesion of disease on CT scan or MRI
* Radiological documentation of disease progression within 12 months prior to randomization
* Adequate liver, renal and bone marrow function
* WHO Performance Status 0-2

Exclusion Criteria:

* Poorly differentiated neuroendocrine carcinoma
* Non-neuroendocrine thymoma
* Patients with severe functional disease who required symptomatic treatment with somatostatin analogs
* Prior therapy with mTOR inhibitors
* History of liver disease
* Baseline QTcF> 470 msec
* Uncontrolled diabetes mellitus despite adequate therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2013-08-16 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (35):
- Denmark (2):
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Copenhagen N
- France (7):
  - Novartis Investigative Site, Toulouse, Cedex 9
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Villejuif
- Germany (3):
  - Novartis Investigative Site, Bad Berka
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Mainz
- Novartis Investigative Site, Athens, GR, Greece
- Italy (10):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Viagrande, CT
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Padua, PD
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Napoli
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Groningen
- Spain (6):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Oviedo, Principality of Asturias
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Lund, Sweden
- United Kingdom (3):
  - Novartis Investigative Site, Withington, Greater Manchester
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on
  https://www.clinicalstudydatarequest.com/

REFERENCES:
- [Derived] Ferolla P, Brizzi MP, Meyer T, Mansoor W, Mazieres J, Do Cao C, Lena H, Berruti A, Damiano V, Buikhuisen W, Gronbaek H, Lombard-Bohas C, Grohe C, Minotti V, Tiseo M, De Castro J, Reed N, Gislimberti G, Singh N, Stankovic M, Oberg K, Baudin E. Efficacy and safety of long-acting pasireotide or everolimus alone or in combination in patients with advanced carcinoids of the lung and thymus (LUNA): an open-label, multicentre, randomised, phase 2 trial. Lancet Oncol. 2017 Dec;18(12):1652-1664. doi: 10.1016/S1470-2045(17)30681-2. Epub 2017 Oct 23. PMID 29074099

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two patients completed the core phase of the study but they did not enter the extension phase one due to worsening in clinical conditions and one for Physician decision.
Period: Core Phase
Arm/Group | Pasireotide LAR | Everolimus | Pasireotide LAR and Everolimus Combination
Started | 41 | 42 | 41
Entered Extension Phase | 12 | 14 | 15
Completed | 12 | 14 | 15
Not Completed | 29 | 28 | 26
Not completed — Adverse Event | 5 | 15 | 13
Not completed — Withdrawal by Subject | 1 | 0 | 3
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Death | 1 | 5 | 2
Not completed — Diseasse progression | 18 | 7 | 8
Not completed — Protocol deviation | 2 | 0 | 0
Not completed — PI decision - did not enter extension | 0 | 1 | 0
Not completed — Worsening of clinical condition - did not enter extension | 1 | 0 | 0
Period: Extension Phase
Arm/Group | Pasireotide LAR | Everolimus | Pasireotide LAR and Everolimus Combination
Started | 12 (Criteria to enter Extension: continued clinical benefit and no unacceptable toxicity) | 14 (Criteria to enter Extension: continued clinical benefit and no unacceptable toxicity) | 15
Completed | 0 | 0 | 0
Not Completed | 12 | 14 | 15
Not completed — Adverse Event | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Administration problems | 3 | 2 | 3
Not completed — Disease progression | 9 | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pasireotide LAR | Everolimus | Pasireotide LAR and Everolimus Combination | Total
Number analyzed (Participants) | 41 | 42 | 41 | 124
Age, Customized [Number; unit: participants]
  18 to <65 | 21 | 18 | 24 | 63
  ≥65 to 84 | 20 | 24 | 17 | 61
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 19 | 13 | 47
  Male | 26 | 23 | 28 | 77
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 40 | 42 | 40 | 122
  Black | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Progression-free at 9 Months Based on Response Evaluation Criteria In Solid Tumors v1.1 (RECIST v1.1)
Description: Patients with Complete Response (CR), Partial Response (PR), or Stable Disease (SD) at Month 9 were to be considered as "progression-free" based on RECIST v1.1. Patients with missing tumor assessment, or with overall lesion response "unknown" at Month 9 were considered as "non progression-free", unless any of the following assessments at Week 48 or Week 52 indicate CR, PR, or SD, in which case the patient was to be considered as progression-free at Month 9. Patients discontinuing the study for any reason prior to the 9 month assessment were to be considered as "non progression-free".
Time Frame: Baseline up to 9 months
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pasireotide LAR | Everolimus | Pasireotide LAR and Everolimus Combination
Number analyzed (Participants) | 41 | 42 | 41
percentage of participants
  Complete response | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 0 [0.0 to 8.6]
  Partial response | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.6] | 2.4 [0.1 to 12.9]
  Stable disease | 34.1 [20.1 to 50.6] | 31.0 [17.6 to 47.1] | 48.8 [32.9 to 64.9]
  Progression-free (PF) at Month 9 | 39.0 [24.2 to 55.5] | 33.3 [19.6 to 49.5] | 58.5 [42.1 to 73.7]

2. Secondary Outcome: Summary of Progression-free Survival (PFS) Based on RECIST v1.1
Description: Time from first study drug administration to objective tumor progression or death from any cause according to RECIST v1.1
Time Frame: Baseline, every 3 months up to 69 months
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pasireotide LAR | Everolimus | Pasireotide LAR and Everolimus Combination
Number analyzed (Participants) | 41 | 42 | 41
months | 8.51 [5.68 to 14.03] | 12.48 [5.55 to 20.21] | 16.53 [11.10 to 23.26]

3. Secondary Outcome: Kaplan-Meier Estimates of Progression-free Survival (PFS)
Description: Percent (%) event-free probability estimate is the estimated probability that a patient will remain event-free up to the specified time point. Percent event-free probability estimates are obtained from the Kaplan-Meier survival estimates. Events are time from first study drug administration to objective tumor progression or death from any cause according to RECIST v1.1.
Time Frame: Baseline, every 3 months up to 69 months
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: event free probability estimates
Arm/Group | Pasireotide LAR | Everolimus | Pasireotide LAR and Everolimus Combination
Number analyzed (Participants) | 41 | 42 | 41
event free probability estimates
  3 months | 83.6 [67.1 to 92.3] | 91.2 [75.1 to 97.1] | 88.6 [72.4 to 95.5]
  6 months | 68.2 [49.8 to 81.1] | 63.5 [44.7 to 77.4] | 85.5 [68.6 to 93.7]
  9 months | 49.6 [31.9 to 65.1] | 56.9 [38.1 to 71.9] | 79.2 [61.1 to 89.5]
  12 months | 39.9 [23.3 to 56.0] | 50.2 [31.9 to 66.0] | 55.5 [36.4 to 71.0]
  15 months | 32.6 [17.2 to 49.1] | 46.8 [28.9 to 62.9] | 51.2 [32.1 to 67.5]
  18 months | 21.8 [9.1 to 37.8] | 38.6 [21.4 to 55.6] | 42.7 [24.2 to 60.1]
  21 months | 14.5 [4.7 to 29.6] | 29.4 [13.6 to 47.2] | 38.0 [20.0 to 55.9]
  24 months | 14.5 [4.7 to 29.6] | 19.6 [6.7 to 37.4] | 28.5 [12.5 to 46.9]
  27 months | 14.5 [4.7 to 29.6] | 19.6 [6.7 to 37.4] | 28.5 [12.5 to 46.9]
  30 months | 10.9 [2.8 to 25.2] | 9.8 [1.8 to 26.2] | 19.0 [6.3 to 36.9]
  33 months | 10.9 [2.8 to 25.2] | 9.8 [1.8 to 26.2] | 19.0 [6.3 to 36.9]
  36 months | 10.9 [2.8 to 25.2] | 9.8 [1.8 to 26.2] | 14.2 [3.7 to 31.5]
  39 months | 10.9 [2.8 to 25.2] | 9.8 [1.8 to 26.2] | 14.2 [3.7 to 31.5]
  42 months | 10.9 [2.8 to 25.2] | 9.8 [1.8 to 26.2] | 14.2 [3.7 to 31.5]
  45 months | 10.9 [2.8 to 25.2] | 9.8 [1.8 to 26.2] | 14.2 [3.7 to 31.5]
  48 months | 10.9 [2.8 to 25.2] | 9.8 [1.8 to 26.2] | 14.2 [3.7 to 31.5]
  51 months | 10.9 [2.8 to 25.2] | NA [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 14.2 [3.7 to 31.5]
  54 months | 10.9 [2.8 to 25.2] | NA [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 14.2 [3.7 to 31.5]
  57 months | 10.9 [2.8 to 25.2] | NA [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 7.1 [0.6 to 25.2]
  60 months | 10.9 [2.8 to 25.2] | NA [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 7.1 [0.6 to 25.2]
  63 months | 10.9 [2.8 to 25.2] | NA [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 7.1 [0.6 to 25.2]
  66 months | NA [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | NA [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 7.1 [0.6 to 25.2]
  69 months | NA [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | NA [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 7.1 [0.6 to 25.2]

4. Secondary Outcome: Summary of Time to Response (Months)
Description: Time from start of treatment to the first observed objective tumor response (partial response or complete response) observed according to RECIST v1.1.
Time Frame: Every 3 months up to Year 1
Population: Full analysis set
Measure: Number; unit: months
Arm/Group | Pasireotide LAR | Everolimus | Pasireotide LAR and Everolimus Combination
Number analyzed (Participants) | 41 | 42 | 41
months
  25th percentile: number analyzed (Participants) | 1 | 1 | 2
  25th percentile | NA — Percentile is not available due to due to insufficient number | NA — Percentile is not available due to due to insufficient number | NA — Percentile is not available due to due to insufficient number
  Median: number analyzed (Participants) | 1 | 1 | 2
  Median | NA — Percentile is not available due to due to insufficient number | NA — Percentile is not available due to due to insufficient number | NA — Percentile is not available due to due to insufficient number
  75th percentile: number analyzed (Participants) | 1 | 1 | 2
  75th percentile | NA — Percentile is not available due to due to insufficient number | NA — Percentile is not available due to due to insufficient number | NA — Percentile is not available due to due to insufficient number

5. Secondary Outcome: Summary of Duration of Response (Months)
Description: Date of first objective tumor response to date of tumor progression or death due to any cause.
Time Frame: Every 3 months up to Year 1
Population: Full analysis set
Measure: Number; unit: months
Arm/Group | Pasireotide LAR | Everolimus | Pasireotide LAR and Everolimus Combination
Number analyzed (Participants) | 41 | 42 | 41
months
  25th percentile: number analyzed (Participants) | 1 | 1 | 2
  25th percentile | NA — Percentile is not available due to due to insufficient number | NA — Percentile is not available due to due to insufficient number | NA — Percentile is not available due to due to insufficient number
  Median: number analyzed (Participants) | 1 | 1 | 2
  Median | NA — Percentile is not available due to due to insufficient number | NA — Percentile is not available due to due to insufficient number | NA — Percentile is not available due to due to insufficient number
  75th percentile: number analyzed (Participants) | 1 | 1 | 2
  75th percentile | NA — Percentile is not available due to due to insufficient number | NA — Percentile is not available due to due to insufficient number | NA — Percentile is not available due to due to insufficient number

6. Secondary Outcome: 12-month Disease Control Rate (DCR) and Objective Response Rate (ORR)
Description: Objective response rate (ORR) was defined as the percentage of patients showing a best overall response (BOR) of CR or PR during the core study according to RECIST v1.1 criteria. The best overall response is interpreted as the best response recorded from the start of the treatment until disease progression/recurrence, death from any cause or until the patient withdraws consent, whichever is earliest. DCR was was defined as the percentage of participants with a best overall response of complete response, partial response or stable disease during 12 months of treatment according to RECIST v1.1.
Time Frame: Baseline up to Month 12
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pasireotide LAR | Everolimus | Pasireotide LAR and Everolimus Combination
Number analyzed (Participants) | 41 | 42 | 41
percentage of participants
  Objective response (CR+PR) | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.6] | 4.9 [0.6 to 16.5]
  Disease control rate (CR+PR+SD) | 80.5 [65.1 to 91.2] | 73.8 [58.0 to 86.1] | 78.0 [62.4 to 89.4]
  Complete response (CR) | 0 [0.0 to 8.6] | 0 [0.0 to 8.4] | 0 [0.0 to 8.6]
  Partial response (PR) | 2.4 [0.1 to 12.9] | 2.4 [0.1 to 12.6] | 4.9 [0.6 to 16.5]
  Stable disease | 78.0 [62.4 to 89.4] | 71.4 [55.4 to 84.3] | 73.2 [57.1 to 85.8]
  Progressive disease | 14.6 [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 4.8 [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 7.3 [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events
  Unknown | 2.4 [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 4.8 [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 0 [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events
  Not assessed | 2.4 [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 16.7 [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 14.6 [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events
  Discontinued before month 12 | 68.3 [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 64.3 [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 63.4 [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events

7. Secondary Outcome: Biochemical Response Rate (BRR) for Chromogranin A (CgA) Levels
Description: Percentage of patients showing normalization or a decrease of ≥ 30% of serum CgA concentrations compared to baseline.
Time Frame: Baseline up to Week 52
Population: Full analysis set participants with CgA levels outside normal range at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pasireotide LAR | Everolimus | Pasireotide LAR and Everolimus Combination
Number analyzed (Participants) | 34 | 27 | 35
percentage of participants
  Week 12 | 20.6 [8.7 to 37.9] | 7.4 [0.9 to 24.3] | 17.1 [6.6 to 33.6]
  Week 24 | 8.8 [1.9 to 23.7] | 7.4 [0.9 to 24.3] | 20.0 [8.4 to 36.9]
  Week 36 | 8.8 [1.9 to 23.7] | 3.7 [0.1 to 19.0] | 11.4 [3.2 to 26.7]
  Week 48 | 8.8 [1.9 to 23.7] | 0 [0.0 to 12.8] | 11.4 [3.2 to 26.7]
  Week 52 | 5.9 [0.7 to 19.7] | 0 [0.0 to 12.8] | 5.7 [0.7 to 19.2]

8. Secondary Outcome: Duration of Biochemical Response (DBR), by Treatment (Full Analysis Set)
Description: Time from the first documentation of biochemical response to the first documentation of biochemical progression or to death due to any cause, whichever occurred first. Biochemical progression is defined as an increase of serum CgA levels ≥ 25% compared to baseline.
Time Frame: Baseline up to Month 18
Population: Full analysis set - participants who have experienced biochemical response during the study and had CgA levels outside normal range at baseline
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pasireotide LAR | Everolimus | Pasireotide LAR and Everolimus Combination
Number analyzed (Participants) | 8 | 4 | 9
months | 14.75 [0.03 to NA] — Upper-bound of CI is non-estimable due to insufficient number of events | 2.00 [0.03 to NA] — Upper-bound of CI is non-estimable due to insufficient number of events | 8.38 [0.03 to NA] — Upper-bound of CI is non-estimable due to insufficient number of events

9. Secondary Outcome: Kaplan-Meier Event-free Probability Estimate Based on CgA Levels
Description: Kaplan Meier estimates are for Duration of biochemical response (DBR) outcome measure. Events are biochemical progressions i.e. an increase of CgA levels >= 25% compared to baseline or deaths due to any cause. Percent (%) Event-free probability estimate is the estimated probability that a patient will remain event-free up to the specified time point.
Time Frame: Baseline, every 3 months up to Month 18
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: event free probability estimates
Arm/Group | Pasireotide LAR | Everolimus | Pasireotide LAR and Everolimus Combination
Number analyzed (Participants) | 8 | 4 | 9
event free probability estimates
  3 months | 75.0 [31.5 to 93.1] | 37.5 [1.1 to 80.8] | 77.8 [36.5 to 93.9]
  6 months | 56.3 [14.7 to 84.2] | NA [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 77.8 [36.5 to 93.9]
  9 months | 56.3 [14.7 to 84.2] | NA [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 44.4 [13.6 to 71.9]
  12 months | 56.3 [14.7 to 84.2] | NA [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 44.4 [13.6 to 71.9]
  15 months | 37.5 [5.6 to 71.7] | NA [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 44.4 [13.6 to 71.9]
  18 months | 37.5 [5.6 to 71.7] | NA [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 44.4 [13.6 to 71.9]

10. Secondary Outcome: Summary of Biochemical Progression-free Survival Based on CgA Levels by Treatment
Description: as for outcome 8
Time Frame: Baseline up Month 24
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pasireotide LAR | Everolimus | Pasireotide LAR and Everolimus Combination
Number analyzed (Participants) | 41 | 42 | 41
months | 2.89 [2.79 to 5.49] | 2.86 [2.79 to 3.52] | 5.62 [3.9 to 8.31]

11. Secondary Outcome: Kaplan-Meier Event-free Probability Estimate for Biochemical Progression-free Survival Based on CgA Levels
Description: Percent (%) Event-free probability estimate is the estimated probability that a patient will remain event-free up to the specified time point. Percent event-free probability estimates are obtained from the Kaplan-Meier survival estimates. Events are biochemical progressions, i.e., an increase of CgA levels >= 25% compared to baseline or deaths due to any cause.
Time Frame: Baseline, every 3 months up to Month 24
Population: Full analysis set
Measure: Number (95% Confidence Interval); unit: event free probability estimates
Arm/Group | Pasireotide LAR | Everolimus | Pasireotide LAR and Everolimus Combination
Number analyzed (Participants) | 41 | 42 | 41
event free probability estimates
  3 months | 43.1 [26.4 to 58.6] | 35.4 [20.0 to 51.1] | 77.1 [59.4 to 87.8]
  6 months | 29.5 [15.0 to 45.6] | 17.7 [7.2 to 32.0] | 44.5 [27.6 to 60.0]
  9 months | 18.5 [7.1 to 34.0] | 11.0 [3.2 to 24.5] | 29.7 [15.5 to 45.2]
  12 months | 18.5 [7.1 to 34.0] | 7.4 [1.4 to 20.0] | 26.4 [13.0 to 41.9]
  15 months | 18.5 [7.1 to 34.0] | NA [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 18.1 [6.7 to 33.8]
  18 months | 13.8 [4.1 to 29.4] | NA [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 18.1 [6.7 to 33.8]
  21 months | 13.8 [4.1 to 29.4] | NA [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 18.1 [6.7 to 33.8]
  24 months | NA [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | NA [NA to NA] — Event-free probability is non-estimable due to insufficient number of participants with events | 18.1 [6.7 to 33.8]

12. Secondary Outcome: Biochemical Response Rate (BRR) for 5HIAA Levels
Description: The percentages are the biochemical response rates i.e. percentage of patients showing normalization i.e. return to within normal ranges, or a decrease of >= 50% from baseline of 5HIAA concentrations.
Time Frame: Baseline up Week 52
Population: Full analysis set - participants with 5HIAA levels within normal range at baseline are excluded from the table, therefore 'n' stands for the number of patients with 5-HIAA levels outside normal range at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Pasireotide LAR | Everolimus | Pasireotide LAR and Everolimus Combination
Number analyzed (Participants) | 20 | 18 | 20
percentage of participants
  Week 12 | 20.0 [5.7 to 43.7] | 11.1 [1.4 to 34.7] | 10.0 [1.2 to 31.7]
  Week 24 | 5.0 [0.1 to 24.9] | 11.1 [1.4 to 34.7] | 20.0 [5.7 to 43.7]
  Week 36 | 5.0 [0.1 to 24.9] | 11.1 [1.4 to 34.7] | 5.0 [0.1 to 24.9]
  Week 48 | 5.0 [0.1 to 24.9] | 0 [0.0 to 18.5] | 5.0 [0.1 to 24.9]
  Week 52 | 5.0 [0.1 to 24.9] | 0 [0.0 to 18.5] | 10.0 [1.2 to 31.7]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 8 weeks post treatment up to maximum duration of 316 weeks
Groups:
- Pasireotide LAR: Pasireotide LAR
- Everolimus: Everolimus
- Pasireotide LAR and Everolimus Combination: Pasireotide LAR and Everolimus Combination
Arm/Group | Pasireotide LAR | Everolimus | Pasireotide LAR and Everolimus Combination
All-Cause Mortality (participants affected / at risk) | 2/41 | 7/42 | 3/41
Serious Adverse Events (participants affected / at risk) | 17/41 | 20/42 | 16/41
Other Adverse Events (participants affected / at risk) | 40/41 | 42/42 | 40/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide LAR (N=41) | Everolimus (N=42) | Pasireotide LAR and Everolimus Combination (N=41)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1 | 0
Tachycardia paroxysmal (Cardiac disorders) | 1 | 0 | 0
Carcinoid crisis (Endocrine disorders) | 0 | 0 | 1
Carcinoid syndrome (Endocrine disorders) | 0 | 1 | 0
Cushing's syndrome (Endocrine disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 2 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Salivary gland pain (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1
Asthenia (General disorders) | 0 | 1 | 0
Axillary pain (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 1
Disease progression (General disorders) | 1 | 1 | 0
Face oedema (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 3 | 2 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 3 | 1
Cholecystocholangitis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0
Aspergillus infection (Infections and infestations) | 0 | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 5 | 2 | 0
Sepsis (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Haematuria traumatic (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperammonaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0
Brain compression (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 2 | 0 | 0
Syncope (Nervous system disorders) | 2 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 1
Anuria (Renal and urinary disorders) | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pasireotide LAR (N=41) | Everolimus (N=42) | Pasireotide LAR and Everolimus Combination (N=41)
Anaemia (Blood and lymphatic system disorders) | 9 | 14 | 10
Leukopenia (Blood and lymphatic system disorders) | 0 | 3 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 9 | 7
Palpitations (Cardiac disorders) | 4 | 1 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 15 | 6 | 6
Abdominal pain upper (Gastrointestinal disorders) | 5 | 5 | 3
Aphthous ulcer (Gastrointestinal disorders) | 0 | 3 | 0
Constipation (Gastrointestinal disorders) | 9 | 6 | 0
Diarrhoea (Gastrointestinal disorders) | 17 | 21 | 33
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 4 | 0
Flatulence (Gastrointestinal disorders) | 2 | 0 | 4
Haemorrhoids (Gastrointestinal disorders) | 3 | 1 | 4
Mouth ulceration (Gastrointestinal disorders) | 0 | 3 | 6
Nausea (Gastrointestinal disorders) | 11 | 10 | 8
Steatorrhoea (Gastrointestinal disorders) | 4 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 2 | 26 | 14
Toothache (Gastrointestinal disorders) | 2 | 1 | 4
Vomiting (Gastrointestinal disorders) | 5 | 5 | 4
Asthenia (General disorders) | 11 | 12 | 16
Chills (General disorders) | 4 | 0 | 0
Fatigue (General disorders) | 6 | 9 | 16
Non-cardiac chest pain (General disorders) | 3 | 4 | 3
Oedema peripheral (General disorders) | 8 | 13 | 12
Pyrexia (General disorders) | 7 | 7 | 6
Bronchitis (Infections and infestations) | 2 | 3 | 1
Cystitis (Infections and infestations) | 1 | 4 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 4
Influenza (Infections and infestations) | 5 | 2 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 4
Rhinitis (Infections and infestations) | 3 | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 2 | 7
Alanine aminotransferase increased (Investigations) | 3 | 3 | 3
Aspartate aminotransferase increased (Investigations) | 4 | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 7 | 2 | 2
Blood creatinine increased (Investigations) | 2 | 1 | 3
Gamma-glutamyltransferase increased (Investigations) | 10 | 4 | 4
Glycosylated haemoglobin increased (Investigations) | 3 | 1 | 3
Platelet count decreased (Investigations) | 0 | 1 | 3
Weight decreased (Investigations) | 18 | 18 | 24
Decreased appetite (Metabolism and nutrition disorders) | 10 | 16 | 13
Diabetes mellitus (Metabolism and nutrition disorders) | 9 | 4 | 8
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 7 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 18 | 14 | 36
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 9 | 5
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 2 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 3 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 3 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 6 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 1 | 4
Dizziness (Nervous system disorders) | 6 | 2 | 2
Dysgeusia (Nervous system disorders) | 4 | 5 | 4
Headache (Nervous system disorders) | 7 | 4 | 6
Presyncope (Nervous system disorders) | 3 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 2 | 4 | 3
Dysuria (Renal and urinary disorders) | 3 | 2 | 1
Polyuria (Renal and urinary disorders) | 1 | 0 | 3
Renal failure (Renal and urinary disorders) | 2 | 4 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 3
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 12 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 11 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 4
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 3 | 3
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2 | 7
Rash (Skin and subcutaneous tissue disorders) | 3 | 12 | 6
Flushing (Vascular disorders) | 1 | 2 | 4
Hypertension (Vascular disorders) | 2 | 2 | 3
Hypotension (Vascular disorders) | 3 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/54/NCT01563354/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT01563354/SAP_001.pdf